CLINICAL TRIAL: NCT05666570
Title: A Study to Demonstrate the Safety and Performance of the Avelle® Negative Pressure Wound Therapy System on Chronic Wounds
Brief Title: The Avelle® Negative Pressure Wound Therapy System on Chronic Wounds
Acronym: SPACE
Status: Withdrawn | Type: Observational
Why Stopped: More cost effective to source real world evidence data
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: WC-22-432
Record Dates: First submitted 2022-09-28; First posted 2022-12-28 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Foot Ulcer; Venous Leg Ulcer
Keywords: negative pressure wound therapy; ulcer
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer; Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Avelle NPWT: Avelle Negative Pressure Wound Therapy administrated as indicated by IFU
  Interventions: Device: Avelle NPWT

INTERVENTIONS:
Device: Avelle NPWT — Wound Management Therapy

SUMMARY:
This study seeks to demonstrate the performance of Negative Pressure Wound Therapy on chronic wounds such as diabetic foot ulcers and venous leg ulcers.

DETAILED DESCRIPTION:
This study seeks to demonstrate the performance of Negative Pressure Wound Therapy on chronic wounds such as diabetic foot ulcers and venous leg ulcers. The primary objective of the study is to demonstrate the performance and safety of Avelle Negative Pressure Wound Therapy on wound and wound fluid management when used in accordance with the instructions for use.

Participation in the study is anticipated to be two weeks. The Avelle™ NPWT System will be used for two weeks and participants will be seen for study visits during this time. Study participants will need to visit the doctor's office up to five times and, at a minimum, will be required to see the health care provider three times, dependent on the condition of the wound. Each visit is anticipated to last for approximately 45 to 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Venous insufficiency as defined by CEAP Classification of C6 or C6R or Diabetic foot ulcer
* Stalled wound/failed treatment in the opinion of the investigator. Defined as a wound that has not progressed by more than 30% in the previous 4 weeks
* 1 qualifying wound which is amenable to NPWT
* Reliable and available for follow-up
* Low to moderate exudate
* Able to tolerate negative pressure
* >18 years old at the time of consent
* Able and willing to provide informed consent

Exclusion Criteria:

* Known sensitivities or allergies to components of the Avelle™ Negative Pressure Wound Therapy System
* Necrotic wounds or wounds with eschar present
* Wound is too small or too large based on wound dressing (> 1cm2 and < 100cm2)
* Wound depth >2cm
* Use of DuoDERM® gel /petroleum gel/ creams/oil-based products
* Active treatment for cancer or completed within the last 3 months
* Severe malnutrition in the opinion of the investigator
* Visible bone/tendon or exposed articular capsule
* Exposed blood vessels
* Clotting disorder
* Malignant wounds
* Systemic infection
* Untreated osteomyelitis
* Patients with HbA1c greater than 9 on Day 0 (Test to be performed within last 3 months)
* Wounds greater than 12 months old
* Previous failed NPWT within last 6 weeks on the qualifying wound
* Active Pregnancy
* Chronic Kidney Disease score of 5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be recruited from the Investigators available population in the anticipated geographies of Colombia and Australia.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-11-27 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
The reduction in wound size of the target wound between baseline and end of study | 14 days
  Area reduction will be assessed by measuring the wound area at Day 0, Day 6 (+/- 1 day), and Day 7 (+/- 1 day)

SECONDARY OUTCOMES:
Wound Healing Status | 14 days
  Assessment of wound progression between baseline and 14 day visit. Wounds will be assessed as healed or progressing towards healing by the investigator.
Assessment of Skin | 14 Days
  Assessment of condition of surrounding skin and signs of infection around the wound using a standardized wound assessment tool (as captured within study database)
Rate of Device Related Adverse Events | 14 days
  Assessment of rate of device related adverse events (ADE) associated with the dressings

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Ulloa, Principal Investigator — Contracted independent health professional
Locations (1):
- Convatec Medical Care, Bogota, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: Undecided